CLINICAL TRIAL: NCT06690086
Title: DERMaSensor Study of Primary Care Physician Use of Elastic-Scattering Spectroscopy (ESS) on Skin Lesions Suggestive of Skin Cancer (DERM-SUCCESS)
Brief Title: DermaSensor Study of Primary Care Physician Use of Elastic-Scattering Spectroscopy (ESS) on Skin Lesions Suggestive of Skin Cancer
Acronym: DERM-SUCCESS
Status: Completed | Type: Observational
Sponsor: DermaSensor, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CSP-18-0002
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Skin Cancer
Keywords: Melanoma; Basal Cell Carcinoma; Squamous Cell Carcinoma; Elastic Scattering Spectroscopy
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with skin lesions suggestive of skin cancer: Subjects with primary skin lesion(s) suggestive of melanoma, basal cell carcinoma, and/or squamous cell carcinoma requiring biopsy to assess the DermaSensor device accuracy in determining risk of malignancy.
  Interventions: Procedure: Lesion biopsy; Device: DermaSensor Device Use

INTERVENTIONS:
Procedure: Lesion biopsy — Lesions enrolled in the study are biopsied to confirm histopathology
Device: DermaSensor Device Use — Users are blinded to the DermaSensor Device result

SUMMARY:
The purpose of this study is to evaluate the clinical validity of the proprietary DermaSensor Elastic Scattering Spectroscopy (ESS) device and classifier algorithm to support assessment of skin lesions suggestive of melanoma, basal cell carcinoma, and/or squamous cell carcinoma in the primary care setting.

DETAILED DESCRIPTION:
A prospective, single-arm, blinded, multicenter study conducted at 22 investigational sites in the United States and Australia. Eighteen sites located in the US and four sites located in Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of any ethnic group aged 22 and older
2. Primary skin lesion suggestive of melanoma, basal cell carcinoma, and/or squamous cell carcinoma that requires biopsy to assess risk of malignancy
3. Patient is willing and able to read, understand and sign the Informed Consent Form (ICF)

Exclusion Criteria:

1. Lesion < 2.5mm in diameter or > 15mm in diameter
2. Lesion surface not accessible (e.g. inside ears, under nails, completely covered by a crust or scale)
3. Lesion on area of crust, psoriasis, eczema or similar skin condition
4. Lesion has erosion and/or ulceration with no area >2.5mm intact
5. Lesion has foreign matter (e.g. tattoo, splinter, dermoscopy oils, or other medicated or non-medicated topical solutions)
6. Lesion in which the device tip cannot be placed entirely within the border of the targeted area
7. Lesion located on acral skin (e.g. sole or palms)
8. Lesion located within 1 cm of the eye
9. Lesion on or adjacent to scars, areas previously biopsied, or areas subjected to any past surgical intervention
10. Lesion located on mucosal surfaces (e.g. genitals, lips)
11. Lesion located on acute sunburn
12. Six (6) or more lesions suggestive of melanoma, basal cell carcinoma, and/or squamous cell carcinoma requiring biopsy to assess risk of malignancy
13. Dementia or other neurologic, physical or psychological limitation that would prevent the patient from signing informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women of any ethnic group aged 22 and older with at least one skin lesion suggestive of melanoma, basal cell carcinoma, and/or squamous cell carcinoma that requires biopsy to assess risk of malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity of DermaSensor for Skin Lesions Suggestive of Melanoma, BCC, and/or SCC | Day 1
Sensitivity + Specificity > 1 for Skin Lesions Suggestive of Melanoma, BCC, and/or SCC | Day 1

SECONDARY OUTCOMES:
Non-inferiority of the DermaSensor sensitivity to the performance goal of 90% | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Merry, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No